CLINICAL TRIAL: NCT01439412
Title: Acupuncture in Acute Nonspecific Low Back Pain; a Randomized Controlled Multicenter Study in General Practice
Brief Title: Acupuncture in Acute Nonspecific Low Back Pain
Acronym: Acuback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Arne Fetveit, Associate Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acuback
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
Keywords: Low back pain; Acupuncture; General practice
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture and standard treatment (Experimental): Adults (20-55 years) who contact their general practitioners office because of acute nonspecific low back pain (0-14 days).
  Interventions: Procedure: Acupuncture and standard treatment
- Standard treatment in general practice (Other): Adults (20-55 years) who contact their general practitioners office because of acute nonspecific low back pain (0-14 days).
  Interventions: Other: Standard treatment in general practice

INTERVENTIONS:
Procedure: Acupuncture and standard treatment — This group will get standard treatment in general practice in accordance with national guidelines, i.e. general advice about activity, prescription of pain relievers (paracetamol, eventually ibuprofen and eventually tramadol), and eventually sick leave.
  In addition they also will receive one treatment of standardized acupuncture procedure during the consultation.
  The acupuncture treatment starts with distal points in the right hand: Lumbar Pain Points (Yaotongxue), strong stimulation for one minute. With the needles still positioned, the patient is instructed to make cautious back and hip movements in 2 minutes. Then the patient lies down on a bench to treat the local points Huatuojiaji ("Jiaji") bilaterally in the segments of the L2-L4 for 5 minutes.
  Other Names: Acupuncture needles:; Seirin B - 8a 0.30 x 30 mm on the Lumbar Pain Points.; Seirin J-8 with sleeve 0.30 x 50 mm on the Jiaji Points.
  Arms: Acupuncture and standard treatment
Other: Standard treatment in general practice — This group will get standard treatment in general practice in accordance with national guidelines, i.e. general advice about activity, prescription of pain relievers (paracetamol, eventually ibuprofen and eventually tramadol), and eventually sick leave.
  Other Names: Standard treatment for low back pain
  Arms: Standard treatment in general practice

SUMMARY:
Acute low back pain is a common disorder in general practice. Some general practitioners (GPs) treat acute low back pain (LBP) with acupuncture, despite lacking evidence of its effectiveness for this condition.

The aim of this study is to evaluate whether a single treatment-session with acupuncture can reduce time to recovery when applied in addition to standard LBP-treatment according to the Norwegian national guidelines. Analyses of prognostic factors for recovery and cost-effectiveness will also be carried out.

The investigators hypotheses are:

1. Acupuncture treatment contributes to faster pain-recovery in acute LBP compared to standard treatment in general practice provided in accordance with the Norwegian national guidelines.
2. Acupuncture treatment for acute LBP improves function, and reduces drug use and sick leave, compared to the standard treatment in general practice provided in accordance with national guidelines.
3. Acupuncture treatment for acute LBP is a cost-effective treatment in general practice.

The investigators intend to include a total of 270 patients, 135 in the intervention group and 135 in the control group.

The investigators planned to do an interim analysis when reaching inclusion of 150 patients. However, this might lead to reduced overall significance level, and as a result of slow inclusion rate (by December 2015), the investigators plan to extend the inclusion time with one year and then complete the study in March 2017.

ELIGIBILITY:
Inclusion Criteria:

* Adults (20-55 years) who contact their general practitioners office because of acute nonspecific low back pain (0-14 days).

Exclusion Criteria:

* Nerve root affection and/or radiating pain below the knee.
* Low back pain with suspected "red flags", i.e. infections, tumors and metastatic disease, rheumatic disease, fractures and significant deformities of the spine.
* Low back pain which starts in pregnancy.
* Physician reported sick leave of 14 days or more during the last month before the back pain, for any reason.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2018-03-17 (Actual); Study Completion 2018-03-17 (Actual)

PRIMARY OUTCOMES:
Median time in days to recovery of pain. | 1 year
  The median time in days to recovery of pain is measured at the first day the patient scores 0 or 1 point on the Numerical Rating Scale (NRS).

SECONDARY OUTCOMES:
Reduction in pain | 1 year
  Pain as measured by the Numeric Rating Scale (NRS), before and immediately after treatment and at the other follow-up times.
Global measure of improvement | 1 year
  Measuring the patients perception of change, stated in whole numbers from 1 = much better to 5 = much worse (Likert improvement scale).
Back specific functional status | 1 year
  Measuring patients' perception of function. The patient answers yes or no concerning 24 allegations about the activities and condition, depending on whether they feel that the statement describes them on this day. Roland Morris Disability Questionnaire.
Sick leaves | 1 year
  The number of days away from work due to back pain.
Use of medication | 1 year
  Use of medication. Paracetamol, eventually others. Counting of daily consumption.
Visits at the GP | 1 year
  Number of new visits at the GP for the back pain.
Side effects of treatment | 1 year
  Reporting of possible side effects of the treatment, both acupuncture and medication.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Fetveit, Dr. Med, Principal Investigator — General Practice Research Unit, Institute of Health and Society, Faculty of Medicine, University of Oslo
Locations (1):
- Institute of Health and Society, Faculty of Medicine, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Skonnord T, Skjeie H, Brekke M, Grotle M, Lund I, Fetveit A. Acupuncture for acute non-specific low back pain: a protocol for a randomised, controlled multicentre intervention study in general practice--the Acuback Study. BMJ Open. 2012 Jun 25;2(3):e001164. doi: 10.1136/bmjopen-2012-001164. Print 2012. PMID 22734119
- [Background] Skonnord T, Skjeie H, Brekke M, Klovning A, Grotle M, Aas E, Mdala I, Fetveit A. Acupuncture for acute non-specific low back pain: a randomised, controlled, multicentre intervention study in general practice-the Acuback study. BMJ Open. 2020 Aug 6;10(8):e034157. doi: 10.1136/bmjopen-2019-034157. PMID 32764081
- [Derived] Skonnord T, Fetveit A, Skjeie H, Brekke M, Grotle M, Klovning A, Aas E. Cost-effectiveness analysis of acupuncture compared with usual care for acute non-specific low back pain: secondary analysis of a randomised controlled trial. Acupunct Med. 2022 Apr;40(2):123-132. doi: 10.1177/09645284211055747. Epub 2021 Nov 30. PMID 34847780